CLINICAL TRIAL: NCT00028301
Title: A Randomized Open-label Study of the Antiviral Efficacy and Safety of Atazanavir Versus Lopinavir/Ritonavir(LPV/RTV), Each in Combination With Two Nucleosides in Subjects Who Have Experienced Virologic Failure With Prior Protease Inhibitor-Containing HAART Regimen(s)
Brief Title: Atazanavir Versus Lopinavir/Ritonavir (LPV/RTV) in Patients Who Have Not Had Success With Protease Inhibitor-Containing HAART Regimen(s)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 302D; AI424-043
Record Dates: First submitted 2001-12-20; First posted 2001-12-21 (Estimated); Last update posted 2010-09-13 (Estimated); Status verified 2010-09

CONDITIONS: HIV Infections
Keywords: HIV Protease Inhibitors; RNA, Viral; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load; Lipids; ABT 378; Antiretroviral Therapy, Highly Active; Lipoproteins, LDL Cholesterol
MeSH Terms: conditions — HIV Infections | interventions — Atazanavir Sulfate; Lopinavir

INTERVENTIONS:
Drug: Atazanavir
Drug: Lopinavir/Ritonavir

SUMMARY:
This study will compare 2 treatments in the way they affect cholesterol levels and the amount of HIV in the blood.

DETAILED DESCRIPTION:
The study is designed to determine the metabolic changes, antiviral activity, safety, and tolerability of atazanavir as compared to LPV/RTV, each in combination with 2 nucleosides, over the initial 24 weeks, with a final analysis at 48 weeks.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are receiving a PI-containing highly active antiretroviral therapy (HAART) for at least 12 weeks.
* Have a viral load of 1,000 or more copies/ml within 4 weeks of screening and within 4 weeks prior to randomization.
* Have 2 CD4 cell counts of 50 or more cells/mm3 at least 96 hours apart and within 4 weeks before randomization.
* Are at least 16 years old.
* Have a documented virologic response to at least 1 HAART regimen.
* Have phenotypic sensitivity to at least 2 of the following: ddl, d4T, ZDV, 3TC, ABC.
* Have phenotypic sensitivity to atazanavir and LPV/RTV.
* Use effective barrier methods of birth control.
* Will be available for 48 weeks.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have taken 2 or more PIs and had virologic failure.
* Have taken atazanavir or LPV/RTV.
* Have an HIV-related infection (within 30 days) or any medical condition requiring treatment at the time of enrollment.
* Have had acute hepatitis in the 30 days prior to study entry.
* Have received certain drugs within 3 months of study start or expect to need them at time of enrollment.
* Abuse alcohol or drugs in a way that would interfere with the study.
* Have very bad diarrhea within 30 days prior to study entry.
* Are pregnant or breast-feeding.
* Have a history of hemophilia.
* Use lipid-lowering drugs (within the previous 30 days).
* Have cardiomyopathy or symptoms of other heart disease.
* Cannot take medicine by mouth.
* Have any other condition that would interfere with the study.
* Have pancreatitis, if choosing ddI as part of NRTI pair.
* Have bilateral peripheral neuropathy at time of screening, if choosing ddI or or d4T as part of the NRTI pair.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-02; Primary Completion 2003-09 (Actual); Study Completion 2003-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (97):
- United States (38):
  - Cooper Green Hosp, Birmingham, Alabama
  - Phoenix Body Positive, Phoenix, Arizona
  - East Bay AIDS Ctr, Berkeley, California
  - Saint Francis Mem Hosp / HIV Care Unit, San Francisco, California
  - Kaiser Foundation Hospital, San Francisco, California
  - San Francisco Veterans Administration Med Ctr, San Francisco, California
  - Harbor UCLA Med Ctr, Torrance, California
  - Beacon Clinic / Boulder Community Hosp, Boulder, Colorado
  - IDC Research Initiative, Altamonte Springs, Florida
  - Larry Bush, Atlantis, Florida
  - Community Health Care, Fort Lauderdale, Florida
  - South Beach Medical Associates, Miami Beach, Florida
  - Florida ID Group, Orlando, Florida
  - Infectious Disease Specialists of Atlanta, Decatur, Georgia
  - Univ of Hawaii, Honolulu, Hawaii
  - Sky Blue, Boise, Idaho
  - Infectious Disease of Indiana, Indianapolis, Indiana
  - Univ of Kansas School of Medicine, Wichita, Kansas
  - Univ of Kentucky Med Ctr, Lexington, Kentucky
  - Community Research Initiative, Brookline, Massachusetts
  - Univ of Massachusetts, Worcester, Massachusetts
  - Southampton Healthcare Inc, St Louis, Missouri
  - Steven Zell, Reno, Nevada
  - VAMC New Jersey Healthcare System, East Orange, New Jersey
  - North Jersey Community Research Initiative, Newark, New Jersey
  - Albany Med College, Albany, New York
  - Erie County Med Ctr, Buffalo, New York
  - North Shore Univ Hosp, Manhasset, New York
  - Community Health Network, Rochester, New York
  - Jemsek Clinic, Huntersville, North Carolina
  - Oregon Health Sciences Univ, Portland, Oregon
  - Research & Education Group, Portland, Oregon
  - Mark Watkins, Philadelphia, Pennsylvania
  - Univ of South Carolina School of Medicine, Columbia, South Carolina
  - North Texas Center for AIDS & Clinical Research, Dallas, Texas
  - Nicholas Bellos, Dallas, Texas
  - Houston Clinical Research Network, Houston, Texas
  - Infectious Diseases Associates of Houston, Houston, Texas
- Argentina (5):
  - Claudia Rodriguez MD, Buenos Aires
  - Elida Pallone MD, Buenos Aires
  - Fundacion Huesped, Buenos Aires
  - Hospital Italiano, Buenos Aires
  - CAICI, Rosario Santa Fe
- Australia (4):
  - Alfred Hosp, Prahan
  - Prahran Market Clinic, South Yarra
  - Saint Vincent's Hosp Med Centre, Sydney
  - Taylors Square Clinic, Sydney
- Belgium (5):
  - Inst of Tropical Medicine, Antwerp
  - CHU Saint Pierre, Brussels
  - Cliniques Universitaires Saint Luc, Brussels
  - University Hospital Gent, Ghent
  - Domaine Universitaire Du SART-TILMAN, Liège
- Brazil (3):
  - Hospital de Clinicas da Universidade Federal do Parana, Curitiba
  - Hospital Nossa Senhora da Conceicao-GCH, Porto Alegre
  - Instituto de Infectologia Emilio Ribas, São Paulo
- Canada (4):
  - Toronto Hosp, Toronto, Ontario
  - Clinique Medicale du Quartier Latin, Montreal, Quebec
  - Dr Roger P Leblanc, Montreal, Quebec
  - Montreal Gen Hosp / Div of Clin Immuno and Allergy, Montreal, Quebec
- Chile (2):
  - Fundacion Arriaran, Santiago
  - Hosp Sotero de Rio, Santiago
- France (5):
  - Hopital Hotel Dieu de Lyon, Lyon
  - CHU De Bicetre, Paris
  - Hopital Cochin - Port Royal, Paris
  - Services des Maladies Infectieuses, Paris
  - Hopital Gustave Dron, Tourcoing
- Italy (9):
  - Ospedale S Orsola, Bologna
  - Immunoligia Universita Cagliari, Cagliari
  - Reparto di Malattie Infettive, Corso Svizzera
  - Ospedale Luigi Sacco Cargnel, Milan
  - Ospedale S Raffaele, Milan
  - Ospedale degli Infermi, Rimini
  - Cat All Immun Clin, Roma
  - Ospedale Amedeo de Savoia, Torino
  - Ospedale Amedeo di Savoia, Torino
- Mexico (4):
  - Hospital 1 ro de Octubre, Mexico City
  - Hospital General, Mexico City
  - Hospital Regional, Mexico City
  - Instituto Nacional de la Nutricion, Mexico City
- Univ Medical Center Utrecht, CX Utrecht, Netherlands
- Peru (2):
  - Hosp Guillermo Almenara-Medicina 1, Lima
  - Hosp Nacional Cayetano Heredia, Lima
- Puerto Rico (2):
  - San Cristobal Hosp, Coto Laurel, Ponce
  - Clinical Research Puerto Rico Inc, San Juan
- Spain (8):
  - Hosp Clinic, Barcelona
  - Hospital Germans Trias I Pujol, Barcelona
  - Hosp de Basurto / Enfermedades Infecciosas, Bilboa
  - Hosp Reina Sofia, Córdoba
  - Hosp Carlos III, Madrid
  - Hosp Ramon y Cajal, Madris
  - Hosp Nuestra Senora de Covadonga, Oviedo
  - Hosp Virgen Del Rocio, Seville
- United Kingdom (2):
  - Whittal Street Clinic, Birmingham
  - Royal Liverpool Univ Hosp, Liverpool
- Country not given (3):
  - Aurora Hospital
  - Department of Infection & Tropical Medicine
  - Klinicka Chorobzkaznych AM